CLINICAL TRIAL: NCT03076372
Title: A Phase-1 Study Evaluating the Safety, Pharmacology and Preliminary Activity of MM-310 in Patients With Solid Tumors
Brief Title: A Study Evaluating MM-310 in Patients With Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Merrimack Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM-310-01-01-01
Record Dates: First submitted 2017-03-01; First posted 2017-03-10 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Solid Tumors; Urothelial Carcinoma; Gastric Carcinoma; Squamous Cell Carcinoma of the Head and Neck; Ovarian Cancer; Pancreatic Ductal Adenocarcinoma; Prostate Adenocarcinoma; Non-small Cell Lung Cancer; Small Cell Lung Cancer; Triple Negative Breast Cancer; Endometrial Carcinoma; Soft Tissue Sarcoma
Keywords: Cancer; Oncology; Phase I; Gemcitabine; Carboplatin; MM-310; EphA2; Ephrin A2; Solid tumors; urothelial carcinoma; gastric carcinoma; squamous cell carcinoma of the head and neck; ovarian cancer; pancreatic ductal adenocarcinoma; prostate adenocarcinoma; non-small cell lung cancer; small cell lung cancer; triple negative breast cancer; endometrial carcinoma; soft tissue sarcoma; Merrimack
MeSH Terms: conditions — Carcinoma, Transitional Cell; Stomach Neoplasms; Squamous Cell Carcinoma of Head and Neck; Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Triple Negative Breast Neoplasms; Endometrial Neoplasms; Sarcoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MM-310 monotherapy (Experimental): MM-310 will be administered by IV infusion over 90 minutes on the first day of each 21 day cycle.
  Interventions: Drug: MM-310

INTERVENTIONS:
Drug: MM-310 — MM-310

SUMMARY:
MM-310 is a liposomal formulation of a docetaxel prodrug that targets the EphA2 receptor on cancer cells. Docetaxel is an approved chemotherapeutic drug.This study is a Phase 1 open-label study of MM-310 in patients with solid tumors. In the first part of the study, MM-310 will be assessed as a monotherapy until a maximum tolerated dose (MTD) is established. After an MTD of MM-310 as a monotherapy is established, an expansion cohort and MM-310 in combination with other therapies will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Must have one of the following cancers, for which the patient has either received or been intolerant to all therapy known to confer clinical benefit

  * Urothelial carcinoma
  * Gastric/gastroesophageal junction/esophageal carcinoma (G/GEJ/E)
  * Squamous Cell Carcinoma of the Head and neck (SCCHN)
  * Ovarian cancer
  * Pancreatic ductal adenocarcinoma (PDAC)
  * Prostate adenocarcinoma (PAC)
  * Non-small cell lung cancer (NSCLC)
  * Small cell lung cancer (SCLC)
  * Triple negative breast cancer (TNBC)
  * Endometrial carcinoma
  * Soft tissue sarcoma subtypes except GIST, desmoid tumors and pleomorphic rhabdomyosarcoma
* Able to provide informed consent, or have a legal representative able and willing to do so
* ≥ 18 years of age
* Availability of a cancerous lesion amenable to biopsy and willing to undergo a pre-treatment biopsy
* ECOG Performance Status of 0 or 1
* Adequate bone marrow reserve as evidenced by:

  * ANC > 1,500/µl (unsupported by growth factors) and
  * Platelet count > 100,000/µl
  * Hemoglobin > 9 g/dL
* Patients must have adequate coagulation function as evidenced by prothrombin time (PT), activated partial thromboplastin time (aPTT) and international normalized ratio (INR) within normal institutional limits
* Adequate hepatic function as evidenced by:

  * Serum total bilirubin ≤ ULN
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN.
  * Alkaline phosphatase ≤ 2.5 x ULN, unless the elevated alkaline phosphatase is due to bone metastasis.
  * In case alkaline phosphatase is >2.5 x ULN patients are eligible for inclusion if aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 1.5 x ULN
* Adequate renal function as evidenced by a serum/plasma creatinine < 1.5 x ULN
* Recovered from the effects of any prior surgery, radiotherapy or other antineoplastic therapy to CTCAE v4.03 grade 1, baseline or less, except for alopecia
* Women of childbearing potential or fertile men and their partners must be willing to abstain from sexual intercourse or to use an effective form of contraception during the study and for 6 months following the last dose of MM-310.

Exclusion Criteria:

* Prior treatment with docetaxel within 6 months of study enrollment
* Pregnant or lactating
* Treatment with systemic anticoagulation (e.g. warfarin, heparin, low molecular weight heparin, anti-Xa inhibitors, etc.) except aspirin
* Any evidence of hematemesis, melena, hematochezia, ≥ grade 2 hemoptysis, or gross hematuria
* Any history of hereditary bleeding disorders
* Presence of an active infection or with an unexplained fever > 38.5°C during screening visits or on the first scheduled day of dosing, which in the investigator's opinion might compromise the patient's participation in the trial or affect the study outcome. At the discretion of the investigator, patients with tumor fever may be enrolled
* Known CNS metastases
* Known hypersensitivity to the components of MM-310, or docetaxel
* Prior treatment with MM-310
* Received treatment, within 28 days or 5 half-lives, whichever is shorter, prior to the first scheduled day of dosing, with any investigational agents that have not received regulatory approval for any indication or disease state and all prior clinically significant treatment related toxicities have resolved to Grade 1 or baseline
* Received other recent antitumor therapy including any standard chemotherapy or radiation within 14 days (or have not yet recovered from any actual toxicities of the most recent therapy) prior to the first scheduled dose of MM-310
* Received any anti-cancer drug known to have anti-VEGF/VEGFR activity within a period of 5 half-lives of this drug (e.g. 100 days for bevacizumab, 75 days for ramucirumab) prior to the first scheduled dose of MM-310
* Clinically significant cardiac disease, including: NYHA Class III or IV congestive heart failure, unstable angina, acute myocardial infarction within six months of planned first dose, arrhythmia requiring therapy (including torsades de pointes, with the exception of extrasystoles, minor conduction abnormalities, or controlled and well treated chronic atrial fibrillation)
* Patients who are not appropriate candidates for participation in this clinical study for any other reason as deemed by the investigator
* Patients who received organ or allogeneic bone marrow or peripheral blood stem cell transplants
* Chronic use of corticosteroids more than 10mg daily prednisone equivalent during the past 4 weeks prior to planned start of MM-310
* Concomitant use of strong inhibitors of CYP3A
* Patients with peripheral neuropathy of grade 2 or higher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2017-02-22 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of MM-310 monotherapy administered once every 3 weeks in patients with metastatic solid tumors. | 18 months

SECONDARY OUTCOMES:
Serum levels of analytes that comprise MM-310 | 18 months
Adverse event profile using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03 | 18 months
Presence of human anti-human antibodies to MM-310 | 18 months
Objective responses based on RECIST v1.1 or other relevant criteria | 18 months
Disease Control Rate | 18 months
Progression Free Survival | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Vasileios Askoxylakis, MD, PhD, Study Director — Merrimack
Locations (5):
- United States (5):
  - Honor Health, Scottsdale, Arizona
  - University California San Francisco, San Francisco, California
  - Mayo Clinic, Rochester, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang ZR, Tipparaju SK, Kirpotin DB, Pien C, Kornaga T, Noble CO, Koshkaryev A, Tran J, Kamoun WS, Drummond DC. Formulation optimization of an ephrin A2 targeted immunoliposome encapsulating reversibly modified taxane prodrugs. J Control Release. 2019 Sep 28;310:47-57. doi: 10.1016/j.jconrel.2019.08.006. Epub 2019 Aug 7. PMID 31400383